CLINICAL TRIAL: NCT03358407
Title: A Single-centre, Randomized, Double-blind (Sponsor Open), Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK2983559, in Single (in Both Fed and Fasted States) and Repeat Oral Doses in Healthy Participants
Brief Title: GSK2983559 First Time in Human Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to non clinical toxicology findings and reduced safety margins.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205021; 2017-002664-40 (EudraCT Number)
Record Dates: First submitted 2017-11-27; First posted 2017-11-30 (Actual); Results first posted 2020-06-22 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel disease; Pro-drug; Double-blinded; Crossover
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: Cohort 1 (Experimental): Cohort 1 will be 5-way crossover with 5 treatment periods. Subjects will be randomized in the ratio 4:1 to receive either single dose of GSK2983559 or placebo.
  Interventions: Drug: GSK2983559; Drug: Placebo
- Part A: Cohort 2 fasting (Experimental): Cohort 2 will be 4-way crossover design with one additional period of open-label. Subjects will be randomized in the ratio 3:1 to receive either single dose of GSK2983559 or placebo in fasted conditions
  Interventions: Drug: GSK2983559; Drug: Placebo
- Part A: Cohort 2 fed (Experimental): In Cohort 2, treatment period 5 will be open-label period. This open-label period is to determine food effect and subjects will receive GSK2983559 under fed conditions.
  Interventions: Drug: GSK2983559
- Part B (Experimental): Part B is repeat ascending dose sequential period. There will four cohorts (3-6) of 10 healthy subjects. In each cohort subjects will be randomized to receive GSK2983559 or placebo in ratio 4:1. Subjects will receive GSK2983559 or placebo QD and twice daily dose will be decided based upon the pharmacokinetic, safety and tolerability observed in Part A.
  Interventions: Drug: GSK2983559; Drug: Placebo

INTERVENTIONS:
Drug: GSK2983559 — GSK2983559 will be available as oral capsules with dose strength of 2-45 milligram (mg), 100 and 114 mg.
Drug: Placebo — Placebo oral capsules matching GSK2983559 will be available for subjects.
  Arms: Part A: Cohort 1; Part A: Cohort 2 fasting; Part B

SUMMARY:
This study is the first administration of GSK2983559, a selective receptor interacting protein 2 (RIP2) kinase inhibitor, to humans. This will be randomized, double-blinded (sponsor open) and two part study (A and B). Part A of the study is single ascending dose crossover design with two separate cohorts (1 and 2). In Part A, 9 single dose levels will be explored. In Cohort 1, 10 healthy subjects will randomized to receive single oral doses of either GSK2983559 or placebo in a ratio of 4:1 in 5 way cross-over design with 5 treatment periods. In Cohort 2, 8 healthy subjects will be randomized to receive single oral doses of either GSK2983559 or placebo in a ratio of 3:1 in 4 way cross-overs design with 4 treatment periods. In Cohort 2 there will be an additional period (period 5-open label) for assessing GSK2983559 under fed conditions. There will be 48 hours wash-out period between each dose escalation period. Part B is repeat ascending dose sequential group design. It will contain 4 Cohorts of and dosing will be done sequential dosing. Subjects in Part B will receive once daily (QD) dose or twice daily dose (will be decided based upon the pharmacokinetic, safety and tolerability observed in Part A). There will 58 subjects involved in this study. Total duration of Part A will be approximately for 11 Weeks and Part B will be approximately for 15 Weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Volunteers who are overtly healthy as determined by medical evaluation including medical and psychiatric history, physical examination, neurological examination, clinical laboratory tests and cardiac monitoring.
* 3Body weight >= 50 kg (kilogram) and body mass index (BMI) within the range 19-32 kilogram per meter square (kg/m^2) .
* A male subject must agree to use a highly effective contraception during the treatment period and for at least 5 half-lives plus an additional 90 days after the last dose of study treatment and refrain from donating sperm during this period.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, and is not a woman of childbearing potential (WOCBP)
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Participants must agree to avoid prolonged Ultraviolet (UV) exposure to natural sunlight without required Ultraviolet A (UVA)/ Ultraviolet B (UVB) protection or tanning beds for the duration of the study.

Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* History or current evidence of febrile seizures, epilepsy, convulsions, significant head injury, or other significant neurologic conditions.
* History of clinically significant psychiatric disorders as judged by the investigator.
* Any history of suicidal behavior within the past 6 months or any history of attempted suicide in a subject's lifetime.
* ALT >1.5x upper limit of normal (ULN).
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of Gastrointestinal (GI) surgery (with exception of appendectomy)
* Average QTc > 450 millisecond (msec)
* Intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to dosing
* Live or attenuated vaccine(s) within 30 days of randomization, or plans to receive such vaccines during the study or plans to receive a vaccine within 30 days + 5 half-lives of the last dose of study medication.
* Regular alcohol consumption within 6 months prior to the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half pint (approximately 240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Current use or history of regular tobacco- or nicotine-containing products within 6 months prior to screening. Subject must have urinary cotinine levels indicative of non-smoking status at screening visit.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrollment or past participation within the last 30 days before signing of consent in this or any other clinical study involving an investigational study treatment or any other type of medical research.
* Subjects with impaired renal function defined as Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) calculation <= 60 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) estimated by the CKD-EPI equation.
* An elevated C-reactive protein (CRP) outside of the normal reference range.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. As potential for and magnitude of immunosuppression with this compound is unknown, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded. Subjects positive for HBsAg and/or positive for anti-HBc antibody (regardless of anti-HBs antibody status) are excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* A positive diagnostic TB test at screening defined as a positive QuantiFERON-TB Gold test or T-spot test. In cases where the QuantiFERON or T-spot test is indeterminate, the subject may have the test repeated once, but they will not be eligible for the study unless the second test is negative. In cases where the QuantiFERON or T-spot test is positive, but a locally-read follow up chest x-ray, shows no evidence of current or previous pulmonary tuberculosis, the subject may be eligible for the study at the discretion of the Investigator and GSK Medical Monitor.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates participation in the study.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Part A (Food Effect) Cohort: Subject must have no dietary restrictions (e.g., lactose intolerance) or inability to eat a high fat meal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of GSK2983559 in healthy participants. The study was terminated early due to non-clinical toxicology findings and reduced safety margins. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Pre-assignment Details: A total of 85 participants were screened, of them, 54 participants were screen failures and 31 participants were enrolled and received study treatment in Part A. The study was terminated during Cohort 2 of Part A, hence no participants were enrolled in period 3, 4 and 5 (Cohort 2) of Part A and in Part B.
Groups:
- Part A-Cohort 1: Placebo/GSK 4mg/GSK 10mg/GSK 30mg/GSK 100mg: Participants (Par.) received oral single dose of placebo matching GSK2983559 (GSK) in treatment period 1 followed by 4 milligram (mg) GSK2983559 in treatment period 2 followed by 10 mg GSK2983559 in treatment period 3 followed by 30 mg GSK2983559 in treatment period 4 followed by 100 mg GSK2983559 in treatment period 5. There was a washout period of at least 48-hours between 2 periods. There was a follow up (FU) visit after 14 days of last period.
- Part A-Cohort 1: GSK 2mg/Placebo/GSK 10mg/GSK 30mg/GSK 100mg: Participants received oral single dose of 2 mg GSK2983559 in treatment period 1 followed by placebo matching GSK2983559 in treatment period 2 followed by 10 mg GSK2983559 in treatment period 3 followed by 30 mg GSK2983559 in treatment period 4 followed by 100 mg GSK2983559 in treatment period 5. There was a washout period of at least 48-hours between 2 periods. There was a follow up visit after 14 days of last period.
- Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg: Participants received oral single dose of 2 mg GSK2983559 in treatment period 1 followed by 4 mg GSK2983559 in treatment period 2 followed by placebo matching GSK2983559 in treatment period 3 followed by 30 mg GSK2983559 in treatment period 4 followed by 100 mg GSK2983559 in treatment period 5. There was a washout period of at least 48-hours between 2 periods. There was a follow up visit after 14 days of last period.
- Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/Placebo/GSK 100mg: Participants received oral single dose of 2 mg GSK2983559 in treatment period 1 followed by 4 mg GSK2983559 in treatment period 2 followed by 10 mg GSK2983559 in treatment period 3 followed by placebo matching GSK2983559 in treatment period 4 followed by 100 mg GSK2983559 in treatment period 5. There was a washout period of at least 48-hours between 2 periods. There was a follow up visit after 14 days of last period.
- Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo: Participants received oral single dose of 2 mg GSK2983559 in treatment period 1 followed by 4 mg GSK2983559 in treatment period 2 followed by 10 mg GSK2983559 in treatment period 3 followed by 30 mg GSK2983559 in treatment period 4 followed by placebo matching GSK2983559 in treatment period 5. There was a washout period of at least 48-hours between 2 periods. There was a follow up visit after 14 days of last period.
- Part A-Cohort 2: Placebo/GSK 400mg: Participants were administered oral single dose of placebo matching GSK2983559 in treatment period 1 followed by 400 mg GSK2983559 in treatment period 2. There was a washout period of at least 48-hours between 2 periods. There was a follow up visit after 14 days of last period. The periods 3, 4, and 5 were planned but no participants were enrolled in those periods due to early terminated of study. The study was terminated during period 2 of Part A-Cohort 2.
- Part A-Cohort 2: GSK 200mg/Placebo: Participants were administered oral single dose of 200 mg GSK2983559 in treatment period 1 followed by placebo matching GSK2983559 in treatment period 2. There was a washout period of at least 48-hours between 2 periods. There was a follow up visit after 14 days of last period. The periods 3, 4, and 5 were planned but no participants were enrolled in those periods due to early terminated of study. The study was terminated during period 2 of Part A-Cohort 2.
- Part A-Cohort 2: GSK 200mg/GSK 400mg: Participants were administered oral single dose of 200 mg GSK2983559 in treatment period 1 followed by 400 mg GSK2983559 in treatment period 2. There was a washout period of at least 48-hours between 2 periods. There was a follow up visit after 14 days of last period. The periods 3, 4, and 5 were planned but no participants were enrolled in those periods due to early terminated of study. The study was terminated during period 2 of Part A-Cohort 2.
- Part B: Placebo: Participants were planned to be administered placebo matching GSK2983559 either once daily or twice daily. Though, no participants were enrolled in Part B since the study was terminated during Part A due to non-clinical toxicology findings and reduced safety margins.
- Part B: GSK2983559: Participants were planned to be administered GSK2983559 in repeat ascending dose sequential period either once daily or twice daily based upon the pharmacokinetic, safety and tolerability observed in Part A. Though, no participants were enrolled in Part B since the study was terminated during Part A due to non-clinical toxicology findings and reduced safety margins.
Period: P1:PartA-Cohort1(4days)+Washout(48hours)
Arm/Group | Part A-Cohort 1: Placebo/GSK 4mg/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/Placebo/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/Placebo/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo | Part A-Cohort 2: Placebo/GSK 400mg | Part A-Cohort 2: GSK 200mg/Placebo | Part A-Cohort 2: GSK 200mg/GSK 400mg | Part B: Placebo | Part B: GSK2983559
Started (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P2:PartA-Cohort1(4days)+Washout(48hours)
Arm/Group | Part A-Cohort 1: Placebo/GSK 4mg/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/Placebo/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/Placebo/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo | Part A-Cohort 2: Placebo/GSK 400mg | Part A-Cohort 2: GSK 200mg/Placebo | Part A-Cohort 2: GSK 200mg/GSK 400mg | Part B: Placebo | Part B: GSK2983559
Started (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P3:PartA-Cohort1(4days)+Washout(48hours)
Arm/Group | Part A-Cohort 1: Placebo/GSK 4mg/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/Placebo/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/Placebo/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo | Part A-Cohort 2: Placebo/GSK 400mg | Part A-Cohort 2: GSK 200mg/Placebo | Part A-Cohort 2: GSK 200mg/GSK 400mg | Part B: Placebo | Part B: GSK2983559
Started (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 2 | 2 | 2 (1 participant was added to Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg arm) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P4:PartA-Cohort1(4days)+Washout(48hours)
Arm/Group | Part A-Cohort 1: Placebo/GSK 4mg/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/Placebo/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/Placebo/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo | Part A-Cohort 2: Placebo/GSK 400mg | Part A-Cohort 2: GSK 200mg/Placebo | Part A-Cohort 2: GSK 200mg/GSK 400mg | Part B: Placebo | Part B: GSK2983559
Started (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: P5:PartA-Cohort1(4days)+Followup(14days)
Arm/Group | Part A-Cohort 1: Placebo/GSK 4mg/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/Placebo/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/Placebo/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo | Part A-Cohort 2: Placebo/GSK 400mg | Part A-Cohort 2: GSK 200mg/Placebo | Part A-Cohort 2: GSK 200mg/GSK 400mg | Part B: Placebo | Part B: GSK2983559
Started (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 2 | 2 | 2 | 2 | 2 (1 participant was added to Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo arm) | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: P1:PartA-Cohort2(4days)+Washout(48hours)
Arm/Group | Part A-Cohort 1: Placebo/GSK 4mg/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/Placebo/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/Placebo/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo | Part A-Cohort 2: Placebo/GSK 400mg | Part A-Cohort 2: GSK 200mg/Placebo | Part A-Cohort 2: GSK 200mg/GSK 400mg | Part B: Placebo | Part B: GSK2983559
Started (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Period: P2:PartA-Cohort2(4days)+Followup(14days)
Arm/Group | Part A-Cohort 1: Placebo/GSK 4mg/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/Placebo/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/Placebo/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo | Part A-Cohort 2: Placebo/GSK 400mg | Part A-Cohort 2: GSK 200mg/Placebo | Part A-Cohort 2: GSK 200mg/GSK 400mg | Part B: Placebo | Part B: GSK2983559
Started (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 0 | 0 | 0 | 0 | 0 | 3 (3 participants were added to Part A-Cohort 2: Placebo/GSK 400mg arm) | 3 (1 participant was added to Part A-Cohort 2: GSK 200mg/ Placebo arm) | 6 (3 participants were added to Part A-Cohort 2: GSK 200mg/GSK 400mg arm) | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 0 | 0
Not completed — Study closed/terminated | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 0 | 0
Period: Part B: Overall Period (11 Weeks)
Arm/Group | Part A-Cohort 1: Placebo/GSK 4mg/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/Placebo/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/Placebo/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo | Part A-Cohort 2: Placebo/GSK 400mg | Part A-Cohort 2: GSK 200mg/Placebo | Part A-Cohort 2: GSK 200mg/GSK 400mg | Part B: Placebo | Part B: GSK2983559
Started (No participants were enrolled in Part B as the study was terminated during Part A.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only data for Part A is presented as study was terminated during Part A and hence Part B was not initiated.
Groups:
- Part A-Cohort 2: GSK 200mg/ Placebo: Participants were administered oral single dose of 200 mg GSK2983559 in treatment period 1 followed by placebo matching GSK2983559 in treatment period 2. There was a washout period of at least 48-hours between 2 periods. There was a follow up visit after 14 days of last period. The periods 3, 4, and 5 were planned but no participants were enrolled in those periods due to early terminated of study. The study was terminated during period 2 of Part A-Cohort 2.
- Total: Total of all reporting groups
Arm/Group | Part A-Cohort 1: Placebo/GSK 4mg/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/Placebo/GSK 10mg/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/Placebo/GSK 30mg/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/Placebo/GSK 100mg | Part A-Cohort 1: GSK 2mg/GSK 4mg/GSK 10mg/GSK 30mg/Placebo | Part A-Cohort 2: Placebo/GSK 400mg | Part A-Cohort 2: GSK 200mg/ Placebo | Part A-Cohort 2: GSK 200mg/GSK 400mg | Part B: Placebo | Part B: GSK2983559 | Total
Number analyzed (Participants) | 2 | 2 | 3 | 2 | 3 | 6 | 4 | 9 | 0 | 0 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] — Only data for Part A is presented as study was terminated during Part A and hence Part B was not initiated.
  Years | 38.0 (11.31) | 46.0 (14.14) | 52.7 (11.85) | 45.5 (13.44) | 59.3 (4.73) | 42.3 (10.50) | 33.8 (7.04) | 42.8 (11.89) |  |  | 44.2 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Only data for Part A is presented as study was terminated during Part A and hence Part B was not initiated.
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Male | 2 | 2 | 3 | 2 | 3 | 6 | 4 | 9 | 0 | 0 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Only data for Part A is presented as study was terminated during Part A and hence Part B was not initiated.
  Participants
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Asian - Central/South Asian Heritage | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3
    White - White/Caucasian/European Heritage | 2 | 2 | 3 | 1 | 3 | 5 | 2 | 9 | 0 | 0 | 27

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Non Serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE was defined as any untoward medical occurrence that, at any dose may result in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement.
Time Frame: Up to 7 weeks
Population: Safety Population comprised of all randomized participants who received at least one dose of study treatment. Data is presented treatment-wise. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Placebo: All participants received single oral dose of placebo matching GSK2983559 as per randomization schedule.
- Part A-Cohort 1: GSK2983559 2 mg: All participants received single oral dose of 2 mg GSK2983559 either in Period 1 or Period 2 or Period 3 or Period 4 or Period 5 as per randomization schedule.
- Part A-Cohort 1: GSK2983559 4 mg: All participants received single oral dose of 4 mg GSK2983559 either in Period 1 or Period 2 or Period 3 or Period 4 or Period 5 as per randomization schedule.
- Part A-Cohort 1: GSK2983559 10 mg: All participants received single oral dose of 10 mg GSK2983559 either in Period 1 or Period 2 or Period 3 or Period 4 or Period 5 as per randomization schedule.
- Part A-Cohort 1: GSK2983559 30 mg: All participants received single oral dose of 30 mg GSK2983559 either in Period 1 or Period 2 or Period 3 or Period 4 or Period 5 as per randomization schedule.
- Part A-Cohort 1: GSK2983559 100 mg: All participants received single oral dose of 100 mg GSK2983559 either in Period 1 or Period 2 or Period 3 or Period 4 or Period 5 as per randomization schedule.
- Part A-Cohort 2: GSK2983559 200 mg: All participants received single oral dose of 200 mg GSK2983559 in Period 1.
- Part A-Cohort 2: GSK2983559 400 mg: All participants received single oral dose of 400 mg GSK2983559 in Period 2.
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Participants
  Non-SAEs | 6 | 2 | 2 | 1 | 1 | 2 | 4 | 4
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Number of Participants With Non-SAEs and SAEs
Description: An adverse event was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE was defined as any untoward medical occurrence that, at any dose may result in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Non-SAEs and SAEs were planned to be collected.
Time Frame: Up to 11 weeks
Population: Safety Population. Data was not collected as no participants were enrolled in Part B due to study termination during Part A.
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Part A: Number of Participants With Worst Case Hematology Parameters of Potential Clinical Importance (PCI)
Description: Hematology parameters included hematocrit, hemoglobin, lymphocytes, platelet counts, total neutrophils and white blood cells (WBCs) count. PCI ranges were: hematocrit (high: >0.54 proportion of red blood cells in blood and low: change from baseline<0.0075); hemoglobin (high: >180 grams per liter [g/L] and low: change from baseline<25 g/L); lymphocytes (low: <0.8 Giga cells/L); platelet count (low: <100 Giga cells/L and high: >550 Giga cells/L); neutrophil count (low: <1.5 Giga cells/L); white blood cell count (low: <3 Giga cells/L and high: >20 Giga cells/L). Participants were counted in the worst-case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category. Only those hematology parameters with PCI values have been presented.
Time Frame: Up to 7 weeks
Population: Safety Population. Data is presented treatment-wise. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Participants
  Hematocrit, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  Hematocrit, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  Hemoglobin, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, To low | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, To within range or no change | 15 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  Lymphocytes, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  Platelet count, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Neutrophils, To low | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Total Neutrophils, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 9
  Total Neutrophils, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC count, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC count, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  WBC count, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part B: Number of Participants With Worst Case Hematology Parameters of PCI
Description: Hematology parameters included hematocrit, hemoglobin, lymphocytes, platelet counts, total neutrophils and WBC count. PCI ranges were: hematocrit (high: >0.54 proportion of red blood cells in blood and low: change from baseline<0.0075); hemoglobin (high: >180 grams per liter [g/L] and low: change from baseline<25 g/L); lymphocytes (low: <0.8 Giga cells/L); platelet count (low: <100 Giga cells/L and high: >550 Giga cells/L); neutrophil count (low: <1.5 Giga cells/L); white blood cell count (low: <3 Giga cells/L and high: >20 Giga cells/L). Participants were counted in the worst-case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category. Participants with worst case hematology parameters of PCI were planned to be collected.
Time Frame: Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Part A: Number of Participants With Worst Case Clinical Chemistry Parameters of PCI
Description: Clinical chemistry parameters included alanine amino transferase (ALT), albumin, alkaline phosphatase (ALP), aspartate amino transferase (AST), calcium, creatinine, glucose, potassium, sodium and total bilirubin (T.bil). PCI ranges were: ALT, AST, ALP (high): >=2*Upper limit of Normal(ULN) units per liter(U/L), albumin(low): 30 g/L, calcium: <2(low) or >2.75 millimoles per liter (mmol/L)(high), creatinine (high): increase from Baseline >44.2 micromoles per liter(µmol/L), glucose: <3(low) or >9 mmol/L(high), potassium: <3(low) or >5.5 mmol/L(high), sodium: <130(low) or >150 mmol/L(high) and T.bil(high): >=1.5*ULN (µmol/L). Participants were counted in the worst case category that their value changes to (low, or within range or no change, or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category.
Time Frame: Up to 7 weeks
Population: Safety Population. Data is presented treatment-wise. Only those clinical chemistry parameters with PCI values have been presented. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Participants
  ALT, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  ALT, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  Albumin, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  ALP, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, To within range or no change | 15 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  AST, To high | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  Calcium, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  Creatinine, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  Glucose, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  Potassium, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  Sodium, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  T.bil, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  T.bil, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  T.bil, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part B: Number of Participants With Worst Case Clinical Chemistry Parameters of PCI
Description: Clinical chemistry parameters included ALT, albumin, alkaline phosphatase, AST, calcium, creatinine, glucose, potassium, sodium and total bilirubin. PCI ranges were ALT(high): >=2*ULN U/L, albumin(low): 30 g/L, alkaline phosphatase(high): >=2*ULN U/L, AST(high): >=2*ULN U/L, calcium: <2(low) or >2.75 mmol/L (high), creatinine (high): increase from Baseline >44.25 µmol/L, glucose: <3(low) or >9 mmol/L(high), potassium: <3(low) or >5.5 mmol/L(high), sodium: <130(low) or >150 mmol/L(high) and total bilirubin(high): >=1.5*ULN (µmol/L). Participants with worst case clinical chemistry parameters of PCI were planned to be collected.
Time Frame: Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Part A: Number of Participants With Worst Case Any Increase in Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method
Description: Urine samples were collected to assess glucose, ketones, occult blood and protein by dipstick method. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters glucose, ketones, occult blood and protein were categorized as 'any increase from Baseline', which imply any increase in their concentrations in the urine sample. Baseline was defined as latest predose (Day 1) assessment with a non-missing value.
Time Frame: Up to 7 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part B: Number of Participants With Worst Case Any Increase in Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method
Description: Urine analysis included assessment of glucose, ketones, occult blood and protein by dipstick method. The dipstick test gives results in a semi-quantitative manner. Baseline was defined as latest predose (Day 1) assessment with a non-missing value. Participants with worst case any increase in urinalysis results post-Baseline relative to Baseline were planned to be collected.
Time Frame: Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Part A: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: 12-lead ECGs were obtained using an ECG machine. Only those participants who had any abnormal ECG findings are presented. Abnormal ECG findings were categorized as clinically significant (CS) and not clinically significant (NCS) abnormal ECG findings. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: 1.5, 2, 2.5, 3, 4, 5, 8, 12, 24 and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles). Data is presented treatment-wise. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Participants
  Abnormal NCS, 1.5 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Abnormal CS, 1.5 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal NCS, 2 hours, n=16,8,8,8,8,8,9,9 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Abnormal CS, 2 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal NCS, 2.5 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Abnormal CS, 2.5 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal NCS, 3 hours, n=6,0,0,0,0,0,9,9: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0 | 9 | 9
  Abnormal NCS, 3 hours, n=6,0,0,0,0,0,9,9 | 0 |  |  |  |  |  | 1 | 0
  Abnormal CS, 3 hours, n=6,0,0,0,0,0,9,9: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0 | 9 | 9
  Abnormal CS, 3 hours, n=6,0,0,0,0,0,9,9 | 0 |  |  |  |  |  | 0 | 0
  Abnormal NCS, 4 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Abnormal CS, 4 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal NCS, 5 hours, n=6,0,0,0,0,0,9,9: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0 | 9 | 9
  Abnormal NCS, 5 hours, n=6,0,0,0,0,0,9,9 | 0 |  |  |  |  |  | 0 | 2
  Abnormal CS, 5 hours, n=6,0,0,0,0,0,9,9: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0 | 9 | 9
  Abnormal CS, 5 hours, n=6,0,0,0,0,0,9,9 | 0 |  |  |  |  |  | 0 | 0
  Abnormal NCS, 8 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
  Abnormal CS, 8 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal NCS, 12 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal CS, 12 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal NCS, 24 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
  Abnormal CS, 24 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal NCS, 48 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal CS, 48 hours, n=16,8,8,8,8,8,9,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Part B: Number of Participants With Abnormal ECG Findings
Description: 12-lead ECGs were planned to be obtained using an ECG machine. Abnormal ECG findings were categorized as CS and NCS abnormal ECG findings. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Participants with any abnormal ECG findings were planned to be evaluated.
Time Frame: Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Part A: Number of Participants With Worst Case Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) Values of PCI
Description: DBP and SBP were measured in semi-supine position after 5 minutes rest. PCI ranges included DBP: <45 millimeters of mercury (mmHg) (lower) and >100 mmHg (higher) and SBP: <85 mmHg (lower) and >160 mmHg (higher). Participants were counted in the worst case category that their value changes to (low, or within range or no change, or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category.
Time Frame: Up to 7 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Participants
  DBP, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  DBP, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, To within range or no change | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
  SBP, To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Part B: Number of Participants With Worst Case DBP and SBP Values of PCI
Description: DBP and SBP were measured in semi-supine position after 5 minutes rest. PCI ranges included DBP: <45 mmHg (lower) and >100 mmHg (higher) and SBP: <85 mmHg (lower) and >160 mmHg (higher). Participants were counted in the worst case category that their value changes to (low, or within range or no change, or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category. Participants with worst case DBP and SBP values of PCI were planned to be evaluated.
Time Frame: Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Part A: Number of Participants With Worst Case Respiration Rate Values of PCI
Description: Respiration rate was measured in semi-supine position after 5 minutes rest. PCI ranges included <=8 breaths per minute (lower) and >=20 breaths per minute (higher). Participants were counted in the worst case category that their value changes to (low, or within range or no change, or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category.
Time Frame: Up to 7 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Participants
  To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  To within range or no change | 12 | 7 | 6 | 8 | 7 | 7 | 7 | 8
  To high | 4 | 1 | 2 | 0 | 1 | 1 | 2 | 1

14. Primary Outcome: Part B: Number of Participants With Worst Case Respiration Rate Values of PCI
Description: Respiration rate was measured in semi-supine position after 5 minutes rest. PCI ranges included <=8 breaths per minute (lower) and >=20 breaths per minute (higher). Participants were counted in the worst case category that their value changes to (low, or within range or no change, or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category. Participants with worst case respiratory rate values of PCI were planned to be evaluated.
Time Frame: Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Part A: Number of Participants With Worst Case Heart Rate Values of PCI
Description: Heart rate was measured in semi-supine position after 5 minutes rest. PCI ranges included <40 beats per minute (lower) and >110 beats per minute (higher). Participants were counted in the worst case category that their value changes to (low, or within range or no change, or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category.
Time Frame: Up to 7 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Participants
  To low | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  To within range or no change | 16 | 8 | 8 | 8 | 8 | 7 | 8 | 9
  To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Part B: Number of Participants With Worst Case Heart Rate Values of PCI
Description: Heart rate was measured in semi-supine position after 5 minutes rest. PCI ranges included <40 beats per minute (lower) and >110 beats per minute (higher). Participants were counted in the worst case category that their value changes to (low, or within range or no change, or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category. Participants with worst case heart rate values of PCI were planned to be evaluated.
Time Frame: Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

17. Primary Outcome: Part A: Number of Participants With Worst Case Body Temperature Values of PCI
Description: Body temperature was measured in semi-supine position after 5 minutes rest. PCI ranges included <=35.5 degrees Celsius (lower) and >=37.8 degrees Celsius (higher). Participants were counted in the worst case category that their value changes to (low, or within range or no change, or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category.
Time Frame: Up to 7 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Participants
  To low | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  To within range or no change | 15 | 8 | 7 | 8 | 8 | 6 | 8 | 7
  To high | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Part B: Number of Participants With Worst Case Body Temperature Values of PCI
Description: Body temperature was measured in semi-supine position after 5 minutes rest. PCI ranges included <=35.5 degrees Celsius (lower) and >=37.8 degrees Celsius (higher). Participants were counted in the worst case category that their value changes to (low, or within range or no change, or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'To within Range or No Change' category. Participants with worst case body temperature values of PCI were planned to be evaluated.
Time Frame: Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

19. Primary Outcome: Part A: Number of Participants With Abnormal Findings in Physical Examination
Description: Physical examinations included assessment of the skin, cardiovascular, respiratory, and gastrointestinal systems. This analysis was not planned and data was not collected and not captured in the database.
Time Frame: Up to 7 weeks
Population: Safety Population. This analysis was not planned and data was not collected and not captured in the database. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Primary Outcome: Part B: Number of Participants With Abnormal Findings in Physical Examination
Description: Physical examinations included assessment of the skin, cardiovascular, respiratory, and gastrointestinal systems. Data was not collected and not captured in the database.
Time Frame: Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Part A: Change From Baseline in Activated Partial Thromboplastin Time and Prothrombin Time at Indicated Time Points
Description: Blood samples were collected to evaluate activated partial thromboplastin time (APTT) and prothrombin time (PT) at indicated time points. Baseline was defined as latest pre-dose (Day 1) assessment with a non-missing value. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose), 24 and 48 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Data is presented treatment-wise. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Seconds
  APTT, 24 hours, n=16,8,8,7,8,8,9,9: number analyzed (Participants) | 16 | 8 | 8 | 7 | 8 | 8 | 9 | 9
  APTT, 24 hours, n=16,8,8,7,8,8,9,9 | 0.4 (3.35) | 0.8 (1.83) | 2.9 (2.85) | -0.7 (1.80) | 1.0 (1.77) | 1.0 (2.56) | -1.3 (6.10) | -1.2 (2.11)
  APTT, 48 hours, n=16,8,8,8,8,8,8,9: number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 9
  APTT, 48 hours, n=16,8,8,8,8,8,8,9 | 0.5 (2.99) | -0.3 (2.66) | 0.5 (3.07) | 0.8 (2.38) | 0.0 (1.69) | 2.3 (2.71) | -3.0 (6.37) | -2.4 (2.96)
  PT, 24 hours, n=16,8,8,7,8,8,9,9: number analyzed (Participants) | 16 | 8 | 8 | 7 | 8 | 8 | 9 | 9
  PT, 24 hours, n=16,8,8,7,8,8,9,9 | 0.1 (0.62) | 0.3 (0.46) | -0.3 (0.46) | 0.1 (0.69) | -0.1 (0.35) | 0.1 (0.35) | -0.2 (1.48) | 0.0 (0.87)
  PT, 48 hours, n=16,8,8,8,8,8,8,9: number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 9
  PT, 48 hours, n=16,8,8,8,8,8,8,9 | -0.1 (0.34) | 0.0 (0.53) | -0.3 (0.46) | 0.1 (0.64) | -0.1 (0.35) | 0.1 (0.35) | -0.4 (1.51) | 0.1 (0.93)

22. Primary Outcome: Part B: Change From Baseline in Activated Partial Thromboplastin Time and Prothrombin Time at Indicated Time Points
Description: Blood samples were planned to be collected to evaluate PTT and PT at indicated time points. Baseline was defined as latest pre-dose (Day 1) assessment with a non-missing value. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

23. Primary Outcome: Part A: Change From Baseline in International Normalized Ratio at Indicated Time Points
Description: Blood samples were collected to evaluate international normalized ratio at indicated time points. Baseline was defined as latest pre-dose (Day 1) assessment with a non-missing value. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose), 24 and 48 hours
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 9 | 9
Ratio
  24 hours, n=16,8,8,7,8,8,9,9: number analyzed (Participants) | 16 | 8 | 8 | 7 | 8 | 8 | 9 | 9
  24 hours, n=16,8,8,7,8,8,9,9 | 0.001 (0.0496) | 0.010 (0.0278) | -0.005 (0.0404) | -0.019 (0.0430) | -0.002 (0.0282) | 0.017 (0.0354) | -0.028 (0.1204) | -0.019 (0.0752)
  48 hours, n=16,8,8,8,8,8,8,9: number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 9
  48 hours, n=16,8,8,8,8,8,8,9 | -0.018 (0.0248) | 0.013 (0.0345) | -0.021 (0.0356) | -0.009 (0.0405) | -0.024 (0.0233) | 0.020 (0.0293) | -0.035 (0.1165) | -0.020 (0.0738)

24. Primary Outcome: Part B: Change From Baseline in International Normalized Ratio at Indicated Time Points
Description: Blood samples were planned to be collected to evaluate international normalized ratio at indicated time points. Baseline was defined as latest pre-dose (Day 1) assessment with a non-missing value. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and Up to 11 weeks
Population: as for outcome 2
Arm/Group | Part B: Placebo | Part B: GSK2983559
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Part A (Cohort 1): Area Under Plasma Concentration-time Curve (AUC) From Zero Hours to Time of Last Quantifiable Concentration (AUC[0-t]) for GSK2983559
Description: Blood samples were collected to measure AUC(0-t) at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods.
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population comprised of all participants in the safety population who had at least 1 non-missing pharmacokinetic assessment. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8
Hours*nanogram per milliliter | NA (NA) — NA indicates that the data is not available since all the concentration data for all participants were below the limit of quantification. | NA (NA) — NA indicates that the data is not available since all the concentration data for all participants were below the limit of quantification. | NA (NA) — NA indicates AUC(0-t) was not calculated due to less than 20% quantifiable concentrations for all participants. | 1.4088 (38.9) | 7.2488 (63.5)

26. Secondary Outcome: Part A (Cohort 2): AUC(0-t) for GSK2983559
Description: as for outcome 25
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 9 | 9
Hours*nanogram per milliliter | 8.1765 (61.7) | 5.9980 (67.3)

27. Secondary Outcome: Part A (Cohort 1): AUC(0-t) for GSK2668176 (Active Moiety of GSK2983559)
Description: Blood samples were collected to measure AUC(0-t) at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Hours*nanogram per milliliter | 96.7389 (19.3) | 250.6231 (36.3) | 390.3911 (17.5) | 889.6956 (17.2) | 2760.8122 (41.3)

28. Secondary Outcome: Part A (Cohort 2): AUC(0-t) for GSK2668176 (Active Moiety of GSK2983559)
Description: as for outcome 27
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 9 | 9
Hours*nanogram per milliliter | 2608.4326 (59.7) | 2857.1378 (39.9)

29. Secondary Outcome: Part A (Cohort 1): AUC From Time Zero to Infinity (AUC[0-inf]) for GSK2983559
Description: Blood samples were collected to measure AUC(0-inf) at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods.
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Hours*nanogram per milliliter | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification.

30. Secondary Outcome: Part A (Cohort 2): AUC(0-inf) for GSK2983559
Description: as for outcome 29
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 9 | 9
Hours*nanogram per milliliter | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification.

31. Secondary Outcome: Part A (Cohort 1): AUC(0-inf) for GSK2668176 (Active Moiety of GSK2983559)
Description: Blood samples were collected to measure AUC(0-inf) at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Hours*nanogram per milliliter | 104.28 (19.4) | 257.28 (36.0) | 405.39 (16.0) | 911.53 (17.1) | 2860.23 (43.0)

32. Secondary Outcome: Part A (Cohort 2): AUC(0-inf) for GSK2668176 (Active Moiety of GSK2983559)
Description: as for outcome 31
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 9 | 9
Hours*nanogram per milliliter | 2717.46 (57.5) | 2950.11 (38.5)

33. Secondary Outcome: Part A (Cohort 1): Maximum Plasma Concentration (Cmax) for GSK2983559
Description: Blood samples were collected to measure Cmax at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods.
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg
Number analyzed (Participants) | 8 | 8 | 2 | 8 | 8
Nanograms per milliliter | NA (NA) — NA indicates that the data is not available since all the concentration data for all participants were below the limit of quantification. | NA (NA) — NA indicates that the data is not available since all the concentration data for all participants were below the limit of quantification. | 0.2291 (12.4) | 0.4034 (37.3) | 1.1937 (40.2)

34. Secondary Outcome: Part A (Cohort 2): Cmax for GSK2983559
Description: as for outcome 33
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 9 | 9
Nanograms per milliliter | 1.3931 (69.3) | 1.1244 (70.0)

35. Secondary Outcome: Part A (Cohort 1): Cmax for GSK2668176 (Active Moiety of GSK2983559)
Description: Blood samples were collected to measure Cmax at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Nanograms per milliliter | 10.4980 (34.5) | 25.9587 (38.6) | 38.4341 (35.5) | 93.8714 (19.5) | 305.9839 (33.0)

36. Secondary Outcome: Part A (Cohort 2): Cmax for GSK2668176 (Active Moiety of GSK2983559)
Description: as for outcome 35
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 9 | 9
Nanograms per milliliter | 314.2321 (113.3) | 351.0316 (68.9)

37. Secondary Outcome: Part A (Cohort 1): Terminal Elimination Half-life (T1/2) for GSK2983559
Description: Blood samples were collected to measure T1/2 at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods.
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Hours | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification.

38. Secondary Outcome: Part A (Cohort 2): T1/2 for GSK2983559
Description: as for outcome 37
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 9 | 9
Hours | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification.

39. Secondary Outcome: Part A (Cohort 1): T1/2 for GSK2668176 (Active Moiety of GSK2983559)
Description: Blood samples were collected to measure T1/2 at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Hours | 7.044 (33.2) | 8.304 (26.9) | 9.649 (26.9) | 8.717 (23.0) | 9.799 (24.7)

40. Secondary Outcome: Part A (Cohort 2): T1/2 for GSK2668176 (Active Moiety of GSK2983559)
Description: as for outcome 39
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 9 | 9
Hours | 10.480 (20.4) | 9.526 (25.6)

41. Secondary Outcome: Part A (Cohort 1): Time to Cmax (Tmax) for GSK2983559
Description: Blood samples were collected to measure Tmax at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods.
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg
Number analyzed (Participants) | 8 | 8 | 2 | 8 | 8
Hours | NA [NA to NA] — NA indicates that the data is not available since all the concentration data for all participants were below the limit of quantification. | NA [NA to NA] — NA indicates that the data is not available since all the concentration data for all participants were below the limit of quantification. | 4.500 [4.00 to 5.00] | 4.005 [3.00 to 5.01] | 4.000 [3.00 to 4.00]

42. Secondary Outcome: Part A (Cohort 2): Tmax for GSK2983559
Description: as for outcome 41
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 9 | 9
Hours | 3.506 [3.00 to 6.00] | 4.000 [3.00 to 5.00]

43. Secondary Outcome: Part A (Cohort 1): Tmax for GSK2668176 (Active Moiety of GSK2983559)
Description: Blood samples were collected to measure Tmax at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Hours | 3.000 [1.51 to 4.00] | 2.758 [2.00 to 4.00] | 4.006 [2.50 to 5.98] | 4.037 [2.00 to 5.01] | 3.000 [2.00 to 4.00]

44. Secondary Outcome: Part A (Cohort 2): Tmax for GSK2668176 (Active Moiety of GSK2983559)
Description: as for outcome 43
Time Frame: Pre-dose and at 15 and 30 minutes; 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 9 | 9
Hours | 3.083 [2.00 to 4.00] | 3.500 [2.00 to 6.00]

45. Secondary Outcome: Part B: AUC(0-t) for GSK2983559 Following Single Dose on Day 1
Description: Blood samples were planned to be collected to measure AUC(0-t) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in each period
Population: Pharmacokinetic Population. Data was not collected as no participants were enrolled in Part B due to study termination during Part A.
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

46. Secondary Outcome: Part B: AUC(0-t) for GSK2983559 on Day 14
Description: Blood samples were planned to be collected to measure AUC(0-t) at indicated time-points.
Time Frame: Day 14: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

47. Secondary Outcome: Part B: AUC(0-t) for GSK2668176 (Active Moiety of GSK2983559) Following Single Dose on Day 1
Description: Blood samples were planned to be collected to measure AUC(0-t) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

48. Secondary Outcome: Part B: AUC(0-t) for GSK2668176 (Active Moiety of GSK2983559) on Day 14
Description: as for outcome 47
Time Frame: as for outcome 46
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

49. Secondary Outcome: Part B: AUC From 0 Hours to the Time of Next Dosing AUC(0-tau) for GSK2983559 Following Single Dose on Day 1
Description: Blood samples were planned to be collected to measure AUC(0-tau) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

50. Secondary Outcome: Part B: AUC(0-tau) for GSK2983559 on Day 14
Description: Blood samples were planned to be collected to measure AUC(0-tau) at indicated time-points.
Time Frame: as for outcome 46
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

51. Secondary Outcome: Part B: AUC(0-tau) for GSK2668176 (Active Moiety of GSK2983559) Following Single Dose on Day 1
Description: Blood samples were planned to be collected to measure AUC(0-tau) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

52. Secondary Outcome: Part B: AUC(0-tau) for GSK2668176 (Active Moiety of GSK2983559) on Day 14
Description: as for outcome 51
Time Frame: as for outcome 46
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

53. Secondary Outcome: Part B: Cmax for GSK2983559 Following Single Dose on Day 1
Description: Blood samples were planned to be collected to measure Cmax at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

54. Secondary Outcome: Part B: Cmax for GSK2983559 on Day 14
Description: Blood samples were planned to be collected to measure Cmax at indicated time-points.
Time Frame: as for outcome 46
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

55. Secondary Outcome: Part B: Cmax for GSK2668176 (Active Moiety of GSK2983559) Following Single Dose on Day 1
Description: Blood samples were planned to be collected to measure Cmax at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

56. Secondary Outcome: Part B: Cmax for GSK2668176 (Active Moiety of GSK2983559) on Day 14
Description: as for outcome 55
Time Frame: as for outcome 46
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

57. Secondary Outcome: Part B: Tmax for GSK2983559 Following Single Dose on Day 1
Description: Blood samples were planned to be collected to measure Tmax at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

58. Secondary Outcome: Part B: Tmax for GSK2983559 on Day 14
Description: Blood samples were planned to be collected to measure Tmax at indicated time-points.
Time Frame: as for outcome 46
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

59. Secondary Outcome: Part B: Tmax for GSK2668176 (Active Moiety of GSK2983559) Following Single Dose on Day 1
Description: Blood samples were planned to be collected to measure Tmax at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

60. Secondary Outcome: Part B: Tmax for GSK2668176 (Active Moiety of GSK2983559) on Day 14
Description: as for outcome 59
Time Frame: as for outcome 46
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

61. Secondary Outcome: Part B: T1/2 for GSK2983559 Following Single Dose on Day 1
Description: Blood samples were planned to be collected to measure T1/2 at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

62. Secondary Outcome: Part B: T1/2 for GSK2983559 on Day 14
Description: Blood samples were planned to be collected to measure T1/2 at indicated time-points.
Time Frame: as for outcome 46
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

63. Secondary Outcome: Part B: T1/2 for GSK2668176 (Active Moiety of GSK2983559) Following Single Dose on Day 1
Description: Blood samples were planned to be collected to measure T1/2 at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

64. Secondary Outcome: Part B: T1/2 for GSK2668176 (Active Moiety of GSK2983559) on Day 14
Description: as for outcome 63
Time Frame: as for outcome 46
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

65. Secondary Outcome: Part B: Accumulation Ratio of GSK2983559
Description: Blood samples were planned to be collected to measure accumulation ratio at indicated time-points. Accumulation ratio was to be calculated as ratio of AUC(0-tau) at Day 14 to AUC(0-tau) at Day 1.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose; Day 14: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose in each period
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

66. Secondary Outcome: Part B: Accumulation Ratio of GSK2668176 (Active Moiety of GSK2983559)
Description: Blood samples were planned to be collected to measure accumulation ratio at indicated time-points. Accumulation ratio was to be calculated as ratio of AUC(0-tau) at Day 14 to AUC(0-tau) at Day 1. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: as for outcome 65
Population: as for outcome 45
Arm/Group | Part B: GSK2983559
Number analyzed (Participants) | 0

67. Secondary Outcome: Part A (Cohort 2): AUC (0-t) for GSK2983559 in Fasted Condition (Period 4)
Description: Blood samples were planned to be collected to measure AUC(0-t) in fasted condition (Period 4) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 4
Population: Pharmacokinetic Population. Data was not collected as no participants were enrolled in period 4 of cohort 2 of Part A as the study was terminated during period 2 of cohort 2 of Part A.
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

68. Secondary Outcome: Part A (Cohort 2): AUC(0-t) for GSK2983559 in Fed Condition (Period 5)
Description: Blood samples were planned to be collected to measure AUC(0-t) in fed condition (Period 5) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 5
Population: Pharmacokinetic Population. Data was not collected as no participants were enrolled in period 5 of cohort 2 of Part A as the study was terminated during period 2 of cohort 2 of Part A.
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

69. Secondary Outcome: Part A (Cohort 2): AUC(0-t) for GSK2668176 (Active Moiety of GSK2983559) in Fasted Condition (Period 4)
Description: Blood samples were planned to be collected to measure AUC(0-t) in fasted condition (Period 4) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 4
Population: as for outcome 67
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

70. Secondary Outcome: Part A (Cohort 2): AUC(0-t) for GSK2668176 (Active Moiety of GSK2983559) in Fed Condition (Period 5)
Description: Blood samples were planned to be collected to measure AUC(0-t) in fed condition (Period 5) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 5
Population: as for outcome 68
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

71. Secondary Outcome: Part A (Cohort 2): AUC(0-inf) for GSK2983559 in Fasted Condition (Period 4)
Description: Blood samples were planned to be collected to measure AUC(0-inf) in fasted condition (Period 4) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 4
Population: as for outcome 67
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

72. Secondary Outcome: Part A (Cohort 2): AUC(0-inf) for GSK2983559 in Fed Condition (Period 5)
Description: Blood samples were planned to be collected to measure AUC(0-inf) in fed condition (Period 5) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 5
Population: as for outcome 68
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

73. Secondary Outcome: Part A (Cohort 2): AUC(0-inf) for GSK2668176 (Active Moiety of GSK2983559) in Fasted Condition (Period 4)
Description: Blood samples were planned to be collected to measure AUC(0-inf) in fasted condition (Period 4) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 4
Population: as for outcome 67
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

74. Secondary Outcome: Part A (Cohort 2): AUC(0-inf) for GSK2668176 (Active Moiety of GSK2983559) in Fed Condition (Period 5)
Description: Blood samples were planned to be collected to measure AUC(0-inf) in fed condition (Period 5) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 5
Population: as for outcome 68
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

75. Secondary Outcome: Part A (Cohort 2): Cmax for GSK2983559 in Fasted Condition (Period 4)
Description: Blood samples were planned to be collected to measure Cmax in fasted condition (Period 4) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 4
Population: as for outcome 67
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

76. Secondary Outcome: Part A (Cohort 2): Cmax for GSK2983559 in Fed Condition (Period 5)
Description: Blood samples were planned to be collected to measure Cmax in fed condition (Period 5) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 5
Population: as for outcome 68
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

77. Secondary Outcome: Part A (Cohort 2): Cmax for GSK2668176 (Active Moiety of GSK2983559) in Fasted Condition (Period 4)
Description: Blood samples were planned to be collected to measure Cmax in fasted condition (Period 4) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 4
Population: as for outcome 67
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

78. Secondary Outcome: Part A (Cohort 2): Cmax for GSK2668176 (Active Moiety of GSK2983559) in Fed Condition (Period 5)
Description: Blood samples were planned to be collected to measure Cmax in fed condition (Period 5) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 5
Population: as for outcome 68
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

79. Secondary Outcome: Part A (Cohort 2): Tmax for GSK2983559 in Fasted Condition (Period 4)
Description: Blood samples were planned to be collected to measure Tmax in fasted condition (Period 4) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 4
Population: as for outcome 67
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

80. Secondary Outcome: Part A (Cohort 2): Tmax for GSK2983559 in Fed Condition (Period 5)
Description: Blood samples were planned to be collected to measure Tmax in fed condition (Period 5) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 5
Population: as for outcome 68
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

81. Secondary Outcome: Part A (Cohort 2): Tmax for GSK2668176 (Active Moiety of GSK2983559) in Fasted Condition (Period 4)
Description: Blood samples were planned to be collected to measure Tmax in fasted condition (Period 4) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 4
Population: as for outcome 67
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

82. Secondary Outcome: Part A (Cohort 2): Tmax for GSK2668176 (Active Moiety of GSK2983559) in Fed Condition (Period 5)
Description: Blood samples were planned to be collected to measure Tmax in fed condition (Period 5) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 5
Population: as for outcome 68
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

83. Secondary Outcome: Part A (Cohort 2): T1/2 for GSK2983559 in Fasted Condition (Period 4)
Description: Blood samples were planned to be collected to measure T1/2 in fasted condition (Period 4) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 4
Population: as for outcome 67
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

84. Secondary Outcome: Part A (Cohort 2): T1/2 for GSK2983559 in Fed Condition (Period 5)
Description: Blood samples were planned to be collected to measure T1/2 in fed condition (Period 5) at indicated time-points.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 5
Population: as for outcome 68
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

85. Secondary Outcome: Part A (Cohort 2): T1/2 for GSK2668176 (Active Moiety of GSK2983559) in Fasted Condition (Period 4)
Description: Blood samples were planned to be collected to measure T1/2 in fasted condition (Period 4) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 4
Population: as for outcome 67
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

86. Secondary Outcome: Part A (Cohort 2): T1/2 for GSK2668176 (Active Moiety of GSK2983559) in Fed Condition (Period 5)
Description: Blood samples were planned to be collected to measure T1/2 in fed condition (Period 5) at indicated time-points. GSK2668176 is the active moiety of pro-drug GSK2983559.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 hours post-dose in Period 5
Population: as for outcome 68
Arm/Group | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were reported from start of study treatment (Day 1) up to Week 7 for Part A
Description: Non-SAEs and SAEs were reported for Safety Population. Adverse events were presented treatment-wise. Data is presented for Part A only as data was not collected in Part B due to the study was terminated during Part A, and Part B was not initiated. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Arm/Group | Part A: Placebo | Part A-Cohort 1: GSK2983559 2 mg | Part A-Cohort 1: GSK2983559 4 mg | Part A-Cohort 1: GSK2983559 10 mg | Part A-Cohort 1: GSK2983559 30 mg | Part A-Cohort 1: GSK2983559 100 mg | Part A-Cohort 2: GSK2983559 200 mg | Part A-Cohort 2: GSK2983559 400 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 6/16 | 2/8 | 2/8 | 1/8 | 1/8 | 2/8 | 4/9 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=16) | Part A-Cohort 1: GSK2983559 2 mg (N=8) | Part A-Cohort 1: GSK2983559 4 mg (N=8) | Part A-Cohort 1: GSK2983559 10 mg (N=8) | Part A-Cohort 1: GSK2983559 30 mg (N=8) | Part A-Cohort 1: GSK2983559 100 mg (N=8) | Part A-Cohort 2: GSK2983559 200 mg (N=9) | Part A-Cohort 2: GSK2983559 400 mg (N=9)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Capillaritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT03358407/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT03358407/SAP_001.pdf